CLINICAL TRIAL: NCT04643509
Title: Cardiac Output Analysis by Cardiographic Impedance: a Validation Study of the Niccomo Non-invasive Monitor in Post-operative Cardiac Surgery
Brief Title: Validity of Cardiac Output Measurement Using Niccomo Device After Cardiac Surgery
Acronym: Niccomo-Card
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2019/020/OB
Record Dates: First submitted 2020-11-19; First posted 2020-11-25 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-11

CONDITIONS: Shock, Cardiogenic; Surgery; Output, Low Cardiac
MeSH Terms: conditions — Shock, Cardiogenic; Cardiac Output, Low

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cardiac surgery: patients benefiting from pulmonary arterial catheter monitoring after cardiac surgery
  Interventions: Device: Niccomo

INTERVENTIONS:
Device: Niccomo — Niccomo monitoring added to pulmonary arterial catheter monitoring

SUMMARY:
Cardiac surgery is at high risk of low cardiac output syndrome after procedure. Monitoring cardiac function, and especially cardiac output, is important to identify cardiovascular dysfunction and to introduce and adjust optimal therapies. Invasive monitor such as pulmonary arterial catheter or transpulmonary thermodilution provide precise measurements but need an invasive access to arterial and central venous route, with possible complications.

Cardiographic bioimpedencemetry (Niccomo device, Imedex Corp) allows a non invasive measurement of cardiac output and some other parameters of cardiovascular function. Nevertheless, the reliability of this device has been little studied after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 y/o
* Patients benefiting from cardiac surgery AND pulmonary arterial catheter monitoring

Exclusion Criteria:

* Aortic regurgitation grade 3-4
* Uncontrolled Hypertension (MAP > 130 mmHg)
* Circulatory or cardiac assistance
* Active pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients bénéfiting from cardiac surgery and pulmonary arterial catheter at the discretion of the physician
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-12-18 (Actual); Primary Completion 2022-12-18 (Estimated); Study Completion 2022-12-23 (Estimated)

PRIMARY OUTCOMES:
agreement between cardiac outputs measured by Pulmonary Arterial Catheter (PAC) and Niccomo | 48 hours
  Cardiac outputs and systolic ejection volumes are measured at 10 different time-points and agreement between the 2 devices are explored

SECONDARY OUTCOMES:
Systolic Time Ratio | 48 hours
  Niccomo values at 10 different time-points
Pre-ejection Period | 48 hours
  Niccomo values at 10 different time-points
Velocity Index | 48 hours
  Niccomo values at 10 different time-points
Left Ventricular Ratio | 48 hours
  Niccomo values at 10 different time-points

CONTACTS AND LOCATIONS:
Locations (1):
- Rouen University Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: Undecided